CLINICAL TRIAL: NCT02860962
Title: A Double-Blind Placebo-Controlled Trial of Dextromethorphan for Treatment of Major Depressive Disorder
Brief Title: A Trial of Dextromethorphan for Treatment of Major Depressive Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00052508
Record Dates: First submitted 2016-08-05; First posted 2016-08-10 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Dextromethorphan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dextromethorphan (Active Comparator): 2 doses of Dextromethorphan 75mg oral (PO), separated by 4 hours
  Interventions: Drug: Dextromethorphan Hydrobromide
- Placebo (Placebo Comparator): 2 doses of placebo (oral/PO), separated by 4 hours
  Interventions: Drug: Dextromethorphan Hydrobromide

INTERVENTIONS:
Drug: Dextromethorphan Hydrobromide — Dose as a single capsule preparation formulated by the Investigational Drug Service of MUSC specifically for the purposes of this trial.

SUMMARY:
A proof-of-concept study to determine the antidepressant potential of Dextromethorphan for treating depression associated with Major Depressive Disorder in inpatients.

DETAILED DESCRIPTION:
The proposed study is a double-blind, placebo-controlled, fixed-dose randomized clinical trial to evaluate the effects of oral Dextromethorphan on psychiatric inpatients hospitalized with Major Depressive Disorder on self and examiner rated inventories of depression. The primary outcome measures will be change in depression symptoms measured with the examiner-rated Montgomery-Åsberg Depression Rating Scale (MADRS). Secondary outcome measures will be depression/anxiety/mood indices measured with subject and examiner-rated inventories including the Beck Depression Inventory-II (BDI), the State-Trait Anxiety Inventory (STAI), and the Clinical Global Impressions Scale (CGI). These additional scales will be used to more comprehensively capture any effects on mood and thought processes that may be missed or under-represented with the use of fewer metrics. The Montgomery-Åsberg Depression Rating Scale was chosen as the primary tool for measurement of depression in this study because it was originally designed for use by trained clinicians in rating depression severity in the inpatient setting, matching the context of the proposed research environment. In order to minimize bias, the research personnel who complete subject assessments taking place on Day 1 and 2 of the study, and during the follow-up visit will be blinded given that assessments on these days involve the completion of examiner-rated scales (MADRS, CGI). Dr. Brueckner (PI) or Dr. Tolliver (co-PI) will be the clinicians performing all screening, initial phase, and follow-up assessments during the course of the study. Blinding will be maintained by the Investigational Drug Service of Medical University of South Carolina (MUSC). Dosing of Dextromethorphan will delivered as two 75mg doses separated by 4 hours. Because there is no preliminary research involving the use of Dextromethorphan in the intended study population, the choice of a total combined dose 150mg dosage represents a best-estimate extrapolation for achieving an adequate pharmacologic effect, while maintaining subject safety. In a study where dextromethorphan was used to investigate its analgesic properties in subjects with Fibromyalgia, statistically significant pain reduction was achieved at a dose of 90mg, but not 60mg. Pain reduction is likely mediated by effects of Dextromethorphan and its primary metabolite Dextrophan on N-methyl-D-aspartate (NMDA) receptors. Adequate binding at this receptor is specifically sought after in this study, as NMDA-receptor antagonism is also the mechanism theorized to impart its potential as a rapid acting antidepressant (although sigma receptor binding may be significantly important as well). Therefore, it is assumed that a dose of at least 90mg is needed to achieve measurable NMDA-receptor activity, and therefore an antidepressant response.

Although only certain concomitant medication regimens will be allowed during the course of the trial as outlined in detail in the inclusion/exclusion criteria below, it should be noted that subjects on certain antidepressant medications like Sertraline, Venlafaxine, Escitalopram, and Bupropion (to name only a few) will be allowed participate in the trial.

As has been discussed so far, and in the following sections of this protocol, studies involving the use of Dextromethorphan for neurological and psychiatric purposes have largely used Dextromethorphan combined with Quinidine, now available as an FDA-approved treatment for Pseudobulbar Affect as a medication called Nuedexta. The Quinidine component inhibits the metabolism of Dextromethorphan, increasing duration of effect, Dextromethorphan plasma levels, and reducing the formation of active metabolite Dextrophan. The decision was made to use dextromethorphan alone in the study for several reasons. The first reason was to avoid introducing undue cardiovascular risk to study participants. Quinidine is an antiarrhythmic drug that can prolong QT interval (although this effect is usually minimal in doses used to achieve inhibition of Dextromethorphan metabolism). Given that many psychiatric medications can prolong QT interval, it was felt that it would be safer not to use Quinidine component along with Dextromethorphan. Secondly, it was felt prudent to ensure that pharmacologic action of Dextromethorphan was not unduly extended (through metabolism inhibition) to protect against the development of protracted side-effects. Additionally, it is actually the primary metabolite of Dextromethorphan, Dextrophan, which has the most robust NMDA receptor antagonist properties. Because action at this receptor is specifically sought due to its presumed antidepressant properties, development of this metabolite is desired, and would be truncated by use of Quinidine or other inhibitors of Dextromethorphan metabolism (for additional details about Dextromethorphan metabolism, and related considerations, see the subsequent sections).

When a subject has undergone screening outlined in the procedural documentation herein and is enrolled in the study, they will be given Dextromethorphan or placebo as two doses. In this study, the investigators will be using Dextromethorphan Hydrobromide Monohydrate powder supplied by the MUSC Investigational Drug Service that will be compounded as a single-capsule preparation with dextrose filler. The placebo will also be provided by the MUSC Investigational Drug Service and consist of dextrose in a single-capsule preparation. Dextromethorphan or placebo will be administered both times with 8 ounces of water. The 75mg dose of Dextromethorphan or the placebo will be administered twice, with the second dosing occurrence taking place 4 hours after the first. In the event that the study subject were to experience a serious adverse event with the initial dose, or be felt to be at risk for an adverse outcome based on their response to the initial dose, they will not be eligible to receive the second dose, and will be removed from the study. Additionally, if the study subject does not want to receive a second dose at the 4 hour mark, their request will be obliged. In the case that this occurs, the remainder of the assessments will occur as normal, as if they did receive the second dose. There will be no requirements regarding food intake or lack thereof before study drug administration on either dosing occasion. Because the effects of a 75mg dose of Dextromethorphan may be subjectively detectable, subject blinding may be compromised due to the presence of interoceptive cues. To detect the presence of this potential issue, subjects participating in this study will be asked to which treatment group they believe they have been assigned. Depression, anxiety, and mood metrics will be obtained 1 hour before dosing of study drug or placebo, at hour 2-4 after the initial dosing, at hour 6-8 hours (2-4 hours after the second dose is administered at the 4 hour mark), and the following day, 24-36 hours after the initial dose. In order to ensure that subjects participating in this study have very intensive follow-up, they will be required to engage in an follow-up visit that will take place the Thursday or Friday following the initial phase of the study, on an inpatient or outpatient basis depending on whether the study subject is discharged from the hospital or not. The same standardized mood assessments will also be obtained during this follow-up visit. During all of these described encounters, adverse events will be recorded, and if necessary additional care will be rendered. The timing, design, and layout of this study were in part extrapolated from a similar study using single-dose intranasal ketamine to treat depression. The timing of measurements was adjusted (compared to the referenced study) to accommodate the pharmacokinetics of Dextromethorphan, enhance study feasibility in the proposed inpatient setting, and allow for 2 doses to be administered to enhance drug exposure. For example, the first encounter with a subject will take place 2-4 hours post-dosing (and 6-8 hours, which is 2-4 post second dosing), as peak plasma levels of Dextromethorphan are usually achieved at this time. In addition to mood metrics obtained during these encounters, during Day 1/Hour -1, Day 1 /Hour 2-4, Day 1/Hour 4, Day 1 /Hour 6-8, and Day 2 /Hour 24-36 the subject will undergo a physical and neurological assessment to monitor for any evidence of untoward medication effect above and beyond adverse events elicited from a verbal exchange with the study subject, based on initial assessment gathered prior to study drug administration (Day 1/Hour -1). This assessment is described below. In line with prior research involving the use of medications with dissociative properties, the Clinician-Administered Dissociative States Scale will be administered in an effort to capture any dissociative signs or symptoms exhibited or experienced by the study subject.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65
2. Meet Diagnostic and Statistical Manual-IV criteria for current Major Depressive Disorder
3. Be receiving inpatient treatment for an acute depressive episode
4. Have voluntarily hospitalization status
5. Have Patient Health Questionnaire (PHQ-9) score of 10 or greater
6. Able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of the assessment instruments.
7. Must consent to random assignment and be willing to commit to medication treatment and follow-up assessments.
8. Negative Urine Drug Screen and Blood Alcohol Level

Exclusion Criteria:

1. A primary psychiatric diagnosis other than Major Depressive Disorder or presence of psychotic features associated with current or past major depressive episodes
2. History of drug induced mania
3. Diagnosis of substance use disorder, as assessed through electronic chart review, or elucidated during screening process
4. Current use of opioids including tramadol, amphetamines/sympathomimetics, or benzodiazepines, prescription or otherwise
5. Abnormal (out of MUSC reference range) kidney function, or liver function > 3x upper limit of normal as per most recent blood work (in inpatient setting either assessed at time of admission, or during the hospitalization)
6. Known pregnancy or positive urine pregnancy test, or breast-feeding
7. History of hypertension, stroke, heart failure, myocardial infarction, Serotonin Syndrome, pulmonary disease, or any currently uncontrolled medical condition that may adversely affect the conduct of the trial or jeopardize the safety of the subject as assessed by research team and or inpatient treatment team
8. Concomitant use of a Monoamine Oxidase Inhibitor or Linezolid (currently, or within 2 weeks of screening)
9. Concomitant use Fluoxetine, Paroxetine, Quinidine, Cinacalcet, or Ritonavir
10. Concomitant use of Memantine, Amantadine, or Ketamine
11. Greater than one serotonergic antidepressant medication (defined as a Selective Serotonin Reuptake Inhibitor/Serotonin-Norepinephrine Reuptake Inhibitor, Tricyclic Antidepressant, or Mirtazapine)
12. A serotonergic antidepressant (defined as a Selective Serotonin Reuptake Inhibitor/Serotonin-Norepinephrine Reuptake Inhibitor, Tricyclic Antidepressant, or Mirtazapine) medication plus any of the following medications: triptans, ergotamines, metoclopramide, buspirone, trazodone, cyclobenzaprine, lithium, or lorcaserin
13. Allergy to or contraindicated use of Dextromethorphan or its excipients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) | Several assessments over the course of 24-36 hours, and during follow-up visit during the following week
  Examiner-rated scale of depression severity

CONTACTS AND LOCATIONS:
Overall Officials: Sudie E. Back, Ph.D., Study Director — Director of Drug and Alcohol Research Track at the Medical University of South Carolina

IPD SHARING:
Plan to Share IPD: Yes